CLINICAL TRIAL: NCT00877201
Title: Improvement of Accommodation With Anti-Oxidant Supplementation in Visual Display Terminal Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryogoku Eye Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ryogoku6886
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Ocular Accommodation
Keywords: Accommodation; visual display terminal (VDT); antioxidant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CDR2

SUMMARY:
The purpose of this study is to determine the antioxidant supplementation effect on accommodation among visual display terminal (VDT) users.

ELIGIBILITY:
Inclusion Criteria:

* best corrected visual acuity is over 20/20

Exclusion Criteria:

* receiving any medication or supplement that would alter the accommodation status within a week from the commencement of this study
* using multifocal spectacles or contact lenses
* pregnant or lactating mothers
* subjects with a history of drug allergy

Ages: 40 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-03

PRIMARY OUTCOMES:
accommodation changes

CONTACTS AND LOCATIONS:
Locations (1):
- Iidabashi Eye Clinic, Tokyo, Japan

REFERENCES:
- [Derived] Uchino Y, Uchino M, Dogru M, Fukagawa K, Tsubota K. Improvement of accommodation with anti-oxidant supplementation in visual display terminal users. J Nutr Health Aging. 2012 May;16(5):478-81. doi: 10.1007/s12603-012-0059-3. PMID 22555795